CLINICAL TRIAL: NCT03926780
Title: Comparative Study of Oral Anticoagulation in Patients With Left Ventricular Thrombi
Brief Title: Comparative Study of Oral Anticoagulation in Left Ventricular Thrombi
Acronym: No-LVT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Young Investigator Group of Cardiovascular Research (Network)
Responsible Party: Principal Investigator, Abdallah Almaghraby, Senior Registrar of Cardiology and Angiology, The Young Investigator Group of Cardiovascular Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YIG01201903
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Anticoagulants; Increased; Left Ventricular Thrombosis
Keywords: warfarin; rivaroxaban; left ventricular thrombus
MeSH Terms: interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Warfarin (Active Comparator): 38 Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE) will be assigned randomly to receive warfarin by the regular starting dose with follow up of the INR to target (2-3)
  Interventions: Drug: Warfarin Sodium
- Rivaroxaban (Experimental): 38 Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE) will be assigned randomly to receive rivaroxaban in a dose of 20 mg per day
  Interventions: Drug: Rivaroxaban 20 MG

INTERVENTIONS:
Drug: Rivaroxaban 20 MG — 38 Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE) will be assigned randomly to receive rivaroxaban 20 mg per day
  Other Names: Xarelto
  Arms: Rivaroxaban
Drug: Warfarin Sodium — 38 Patients with evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE) will be assigned randomly to receive warfarin sodium by a dose starting from 3 mg per day and titrated accordingly to target an INR of 2-3
  Other Names: Marevan
  Arms: Warfarin

SUMMARY:
Left ventricular (LV) thrombus is a common problem that is encountered in patients who survived from a large myocardial infarction, and distal systemic embolization is the main issue in these patients due to its major clinical consequences especially cerebrovascular stroke.

Novel oral anticoagulants (NOACs) are now used safely in nonvalvular atrial fibrillation, these agents were shown to be at least as effective as Vitamin K antagonists (VKA) such as warfarin in prevention of systemic embolism, while having an improved safety profile with less bleeding risk. However, the data about their usage for LV thrombi instead of the commonly used VKA are still lacking except for case reports and small case series.

The proposed aim of this randomized observational clinical trial is to assess the efficacy of the conventional anticoagulation in the form of warfarin and NOACs in the form of rivaroxaban in the treatment of LV thrombus.

DETAILED DESCRIPTION:
The proposed aim of this randomized observational clinical trial is to assess the efficacy of the conventional anticoagulation in the form of warfarin and NOACs in the form of rivaroxaban in the treatment of LV thrombus.

So patients with actual LV thrombus will be divided into 2 groups, one will receive the traditional therapy which is warfarin with follow up of the INR in order to reach the desired level of 2-3 then follow up every two weeks to determine the time in therapeutic range until the end of the study follow up. The other group will receive oral rivaroxaban 20 mg per day with follow up for the persistence or the disappearance of the LV thrombus one month, three months and 6 months later.

As a secondary and safety end point, any major bleeding will be recorded as well as any thrombo-embolic events

ELIGIBILITY:
Inclusion Criteria:

* Evidence of LV thrombus as assessed by trans-thoracic echocardiography (TTE).

Exclusion Criteria:

* Creatinine clearance less than 50 ml/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Presence or absence of left ventricular thrombus as assessed by 2D transthoracic echocardiography | 1 month
  2D transthoracic echocardiography will be done after 1 month of initiation of the anticoagulant in order to assess the presence/absence of the thrombus
Presence or absence of left ventricular thrombus as assessed by 2D transthoracic echocardiography | 3 months
  2D transthoracic echocardiography will be done after 3 months of initiation of the anticoagulant in order to assess the presence/absence of the thrombus
Presence or absence of left ventricular thrombus as assessed by 2D transthoracic echocardiography | 6 months
  2D transthoracic echocardiography will be done after 6 months of initiation of the anticoagulant in order to assess the presence/absence of the thrombus

SECONDARY OUTCOMES:
Stroke or systemic embolism | Up to 6 months
  Any type of stroke or systemic embolism event will be recorded
Major bleeding | Up to 6 months
  Any major bleeding that may occur according to the criteria of the International Society on Thrombosis and Haemostasis (ISTH) will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Haitham Badran, PhD, Study Director — Assisstant Professor of Cardiology and Angiology, University of Ain Shams, Egypt
Locations (1):
- Andalusia Hospitals, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelnabi M, Saleh Y, Fareed A, Nossikof A, Wang L, Morsi M, Eshak N, Abdelkarim O, Badran H, Almaghraby A. Comparative Study of Oral Anticoagulation in Left Ventricular Thrombi (No-LVT Trial). J Am Coll Cardiol. 2021 Mar 30;77(12):1590-1592. doi: 10.1016/j.jacc.2021.01.049. No abstract available. PMID 33766266